CLINICAL TRIAL: NCT02924948
Title: A Comparison of Endoscopic Ultrasound Insertion Methods: Conventional vs Inflated Balloon Method
Brief Title: A Comparison of Endoscopic Ultrasound Insertion Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0315
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Throat Pain After EUS Insertion
Keywords: Endoscopic ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional insertion (No Intervention): EUS will be inserted with conventional method.
- Balloon inflated insertion (Experimental): EUS will be inserted with balloon inflated method
  Interventions: Procedure: Balloon inflation

INTERVENTIONS:
Procedure: Balloon inflation — EUS balloon inflation will be done before insertion through the subjects throat
  Arms: Balloon inflated insertion

SUMMARY:
Endoscopic ultrasonography (EUS) is an essential technique required in diagnosis of pancreatobiliary diseases. In previous studies, 6% of patients who undergone EUS had significant throat pain. (NRS scale 5 or greater) Although some endoscopists think balloon inflation while EUS insertion could result in decreased throat damage and pain, there is no data to back up. We designed a single center randomized pilot study to compare throat pain caused by EUS insertion with conventional vs balloon inflation method.

DETAILED DESCRIPTION:
All patients who are undergoing EUS with radial type echoendoscope will be asked for an informed consent. Subjects will be randomized to conventional insertion arm and balloon inflated insertion arm. All patients will be sedated according to SNUH endoscopy center protocol. Conventional insertion will be done in conventional insertion group, and balloon inflation before the start of procedure will be done in balloon inflated insertion arm. After the EUS procedure is finished, subject will be moved to a recovery room. As soon as the subject is recovered from sedation, throat pain will be assessed in NRS scale and be recoreded. Information of insertion failure and balloon damage during insertion will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 to 80
* Patients undergoing EUS with radial echoendoscope

Exclusion Criteria:

* Refuse to participate the study
* Refuse EUS procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Throat pain | Assess right after the end of the EUS procedure
  Throat pain assessed by NRS scale 5 or over will be considered as positive

SECONDARY OUTCOMES:
Throat pain intensity | Assess right after the end of the EUS procedure
  Throat pain assessed in NRS scale which has a range of 0 to 10
EUS Insertion failure rate | Right after insertion
  To assess the EUS insertion failure rate
Damaged balloon rate | during EUS procedure
  Inability to inflate the balloon after insertion of EUS will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD. PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No